CLINICAL TRIAL: NCT01055522
Title: Dose Definition and Activity Evaluation Study of the Tumor-Targeting Human L19IL2 Monoclonal Antibody-Cytokine Fusion Protein in Combination With Dacarbazine in Patients With Metastatic Melanoma
Brief Title: Clinical Study Phase II of L19IL2 in Combination With Dacarbazine in Patients With Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Collaborators: Eudax S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19IL2DTIC-03/07; 2007-005737-11 (EudraCT Number)
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2012-10

CONDITIONS: Metastatic Melanoma
Keywords: Interleukin, IL2, monoclonal, antibody, cytokine, Dacarbazine, metastatic, melanoma, tumor targeting, Dose definition; , L19
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ARM 1: L19IL2 + Dacarbazin (Experimental)
  Interventions: Drug: Arm 1: L19IL2 + Dacarbazine
- ARM 2: L19IL2 + Dacarbazin (Experimental)
  Interventions: Drug: ARM 2: L19IL2 + Dacarbazine
- ARM 3: Dacarbazin (Active Comparator): DTIC every three weeks until disease progression, unacceptable toxicity, withdrawal of consent, or for a maximum of 8 cycles, whichever occurs first
  Interventions: Drug: Arm 3: Dacarbazine

INTERVENTIONS:
Drug: Arm 1: L19IL2 + Dacarbazine — RD of L19IL2 determined in phase IIa. Induction Phase A: Intravenous (IV) infusion of L19IL2 on days 1, 3 and 5 of each 21-day cycle over 60 minutes via automated device (perfusor), for four consecutive 21-day cycles.
  Induction Phase B: Intravenous (IV) infusion of L19IL2 on days 1, 8 and 15 of each 21-day cycle over 60 minutes via automated device (perfusor), for four consecutive 21-day cycles.
  Maintenance: Intravenous (IV) infusion of L19IL2 on days 1, 8 and 15 of each 21-day cycle over 60 minutes via automated device (perfusor), for a maximum of 1 year after start of treatment.
  DTIC 1,000mg/m2 every three weeks until disease progression, unacceptable toxicity, withdrawal of consent, or one year from initiation of therapy, whichever occurs first
  Arms: ARM 1: L19IL2 + Dacarbazin
Drug: Arm 3: Dacarbazine — Dacarbazine Dosage: 1,000 mg/m2 DTIC every three weeks until disease progression, unacceptable toxicity, withdrawal of consent, or for a maximum of 8 cycles, whichever occurs first.
  Other Names: DETICENE®
  Arms: ARM 3: Dacarbazin
Drug: ARM 2: L19IL2 + Dacarbazine — RD of L19IL2 determined in phase IIa. Intravenous (IV) infusion of L19IL2 on days 1, 8 and 15 of each 21-day cycle over 60 minutes via automated device (perfusor), for for a maximum of 1 year after start of treatment.
  DTIC 1,000mg/m2 every three weeks until disease progression, unacceptable toxicity, withdrawal of consent, or one year from initiation of therapy, whichever occurs first
  Arms: ARM 2: L19IL2 + Dacarbazin

SUMMARY:
This Phase II clinical study is an open-label, multicenter study of L19IL2 in combination with Dacarbazine in patients with metastatic melanoma.

The study is divided in two parts: a phase IIa part, designed to establish the recommended dose (RD) of L19IL2 when administered in combination with a fixed dose of Dacarbazine, as well as to determine the preliminary tolerability profile; the second phase IIb part evaluates the objective response rate (ORR) including a randomized study with a fixed dose of Dacarbazine with or without L19IL2, dosed at the RD determined in phase IIa.

DETAILED DESCRIPTION:
Dose limiting toxicity will be assessed during the dose-escalation part of Phase IIa from day 1 through day 21 of the first cycle.

Response will be measured using RECIST criteria every 6 weeks (after every 2 cycles of treatment). Patients with stable or responding disease at each assessment may receive additional treatment for a maximum of 6 cycles of induction. Patients with stable or responding disease after induction may receive L19IL2 (without dacarbazine) every 2 weeks as maintenance therapy.

Tumor expression of ED-B FN and tumor uptake of L19IL2 and of Dacarbazine will be assessed via immunohistochemistry and/or other methods deemed appropriate on tumor tissue biopsies. Tumor biopsy will be performed on superficial accessible cutaneous and/or subcutaneous lesions only. Tumor biopsy will be considered optional and will not preclude patient entry on to study should the patient refuse.

Pharmacokinetics of L19IL2, Dacarbazine and AIC will be assessed from serial blood samples using standard methods.

Overall response rate, PFS, survival rate at 6 and 12 months, and overall survival time for all patients and separately for the patients in the Phase IIb part will be assessed using standard methods.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed unresectable metastatic (stage IV) non-uveal melanoma
* Age > 18 years
* Measurable disease defined as at least one lesion that can be accurately and serially measured per the modified RECIST criteria. Cutaneous lesions measuring at least 1 cm will be considered measurable.
* Prior therapy for metastatic melanoma:

  * Phase IIa - Dose definition: prior therapy allowed, including prior chemotherapy; previous treatment with DTIC: patients should be treated > 6 months prior to study entry
  * Phase IIb -Activity Evaluation: no prior therapy except radiation. However, if radiation has been administered to a lesion, there must be radiographic evidence of progression of that lesion in order for that lesion to constitute measurable disease or to be included in the measured target lesions
* Fewer than 3 organs involved or cutaneous and/or subcutaneous metastasis only, for PhaseIIb patients
* ECOG performance status < 2
* Life expectancy of at least 12 weeks
* Absolute neutrophil count > 1.5 x 109/L, hemoglobin > 9.0 g/dL and platelets > 100 x 109/L
* Total bilirubin ≤ 30 µmol/L (or ≤ 2.0 mg/Dl)
* ALT and AST ≤ 2.5 x the upper limit of normal (5.0 x ULN for patients with hepatic involvement with tumor
* LDH < 2.0 x ULN for Phase IIa patients and normal LDH for the Phase IIb ones.
* Serum creatinine < 1.5 x ULN
* All toxic effects of prior therapy must have resolved to ≤ Grade 1 unless otherwise specified above
* Negative serum pregnancy test (for women of child-bearing potential only) at screening

Exclusion criteria:

* Primary ocular melanoma
* Evidence of brain metastases, negative CT scan within two months before study commence
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (TA, Tis & Ti) or any cancer curatively treated < 5 years prior to study entry
* History of HIV infection or chronic hepatitis B or C
* Presence of active infections (e.g. requiring antimicrobial therapy) or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
* Inadequately controlled cardiac arrhythmias including atrial fibrillation
* History within the last year of acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
* Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria).
* Uncontrolled hypertension.
* Ischemic peripheral vascular disease (Grade Iib-IV).
* Severe diabetic retinopathy.
* Active autoimmune disease
* History of organ allograft or stem cell transplantation.
* Recovery from major trauma including surgery within 4 weeks prior to administration of study treatment.
* Known history of allergy to IL2, dacarbazine, or other intravenously administered human proteins/peptides/antibodies.
* Breast feeding female.
* Anti-tumor therapy within 4 weeks of the administration of study treatment.
* Previous in vivo exposure to monoclonal antibodies for biological therapy in the 6 weeks before administration of study treatment.
* Previous DTIC treatment in the last 6 months prior to study entry
* Growth factors or immunomodulatory agents within 7 days of the administration of study treatment.
* Patient requires or is taking corticosteroids or other immunosuppressant drugs on a long-term basis. Limited use of corticosteroids to treat or prevent acute hypersensitivity reactions is not considered an exclusion criterion.
* Any conditions that in the opinion of the investigator could hamper compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2008-06; Primary Completion 2013-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To establish the recommended dose (RD) of L19IL2 when administered in combination with a fixed dose of Dacarbazine | 21 days
To evaluate Objective response rate (ORR) by CT or MRI | 18 weeks

SECONDARY OUTCOMES:
To investigate the Pharmacokinetics of L19IL2, dacarbazine and 5-aminoimidazole -4 carboxamide (AIC). | 42 days
To investigate the induction of human anti-fusion protein antibodies (HAFA) | 1 year
To investigate Antitumor activity of L19IL2 with dacarbazine in patients with metastatic melanoma by TC or MRI | 18 weeks
Evaluation of the immunological activity of study treatment | 1 year
To estimate progression -free survival (PFS) | 1 year
To estimate overall survival (OS) | 1 year
To assess safety and tolerability | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Matilde Catania, Dr, Principal Investigator — European Istitute of Oncology Milan (Italy); Claus Garbe, Prof. M.D., Principal Investigator — University Hospital Tuebingen (Germany)
Locations (10):
- Universitätsklinik Graz, Graz, Austria
- Germany (3):
  - Charité- Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Schleswig-Holstein-Campus Kiel, Kiel
  - University Hospital, Tübingen
- Italy (5):
  - University Hospital Pisa, Pisa, Tuscany
  - A.O. UNIVERSITARIA OSPEDALI RIUNITI - OSPEDALE UMBERTO I DI ANCONA - ANCONA (AN) (Italy), Ancona
  - European Institute of Oncology, Milan
  - Istituto Nazionale Per Lo Studio E La Cura Dei Tumori Fondazione Giovanni Pascale Di Napoli, Napoli
  - Azienda Ospedaliera Universitaria Senese, Siena
- Universitäts Spital Zürich, Zurich, Switzerland

REFERENCES:
- [Derived] Eigentler TK, Weide B, de Braud F, Spitaleri G, Romanini A, Pflugfelder A, Gonzalez-Iglesias R, Tasciotti A, Giovannoni L, Schwager K, Lovato V, Kaspar M, Trachsel E, Menssen HD, Neri D, Garbe C. A dose-escalation and signal-generating study of the immunocytokine L19-IL2 in combination with dacarbazine for the therapy of patients with metastatic melanoma. Clin Cancer Res. 2011 Dec 15;17(24):7732-42. doi: 10.1158/1078-0432.CCR-11-1203. Epub 2011 Oct 25. PMID 22028492